CLINICAL TRIAL: NCT05246761
Title: To Study the Effectiveness and Safety of Balloon Catheter Combined With Oxytocin Induction Among the Pregnant Women With Previous Cesarean Section: Multicenter, Prospective, Observational Study
Brief Title: Balloon Catheter Combined With Oxytocin Induction Among the Pregnant Women With Previous Cesarean Section
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: JPPTOLAC-01
Record Dates: First submitted 2022-01-13; First posted 2022-02-18 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Trial of Labor After Cesarean; Vaginal Birth After Cesarean; Bishop Score; Failed Mechanical Induction; Balloon Catheter for Labor Induction; Unfavorable Cervix

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cesarean section group: In the cesarean section group, all the pregnant women had only one prior cesarean section.
  Interventions: Device: Balloon catheter
- Non-cesarean section group: In the non-cesarean section group, all the pregnant women are primipara，and never had a cesarean section.
  Interventions: Device: Balloon catheter

INTERVENTIONS:
Device: Balloon catheter — In the two groups, if their bishop score <6, they will receive the cervical riening by the balloon catheter, and then the oxytocin if necessary.

SUMMARY:
This study is a multi-center, prospective, observational clinical trial study. 924 full-term pregnant women will be enrolled as subjects, and the ratio of eligible subjects in the two groups is 1:1. In the prior cesarean section group, pregnant women with one previous cesarean section who are willing to try to the trial of labor after cesarean (TOLAC) and in accordance with the criteria according to the 2016 China vaginal birth after cesarean (VBAC) clinical management guidelines will be enrolled and recorded by our homemade registration form of TOLAC. In the control group, pregnant women after 39 weeks of gestation without vaginal labor contraindications will be enrolled. Whether in the experimental group or the control group, their cervical bishop score was less than 6 points, and they all will be induced by balloon catheter + oxytocin. After 96h, their final delivery mode will be recorded. In the following 42 days postpartum, their complications and the neonatal outcome will be followed up.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers sign the informed consent;
2. Age: 20-40 years;
3. Singleton, a cephalic presentation;
4. No contradiction to vaginal delivery; 5.39~42 weeks.

Exclusion criteria:

1. Konwn contraindication to vaginal delivery or severe complications;
2. Multiple gestation;
3. Uterine malformation;
4. Severe psychiatric disorder;
5. Without family's support.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: In the cesarean section group, the extra inclusion criteria includes:
  Only one prior low transverse uterine incision;
  Extra exclusion criteria:
  1. With mutiple history of c esction;
  2. Prior extensive transfundal uterine surgery, such as for fetal surgery, myomectomy, or uterine reconstruction; Prior classical vertical uterine incision, or an inverted "T" or "J" incision;
  3. Short interpregnancy interval;
  4. Prior uterine rupture or dehiscence, or cesarean scar pregnancy;
  5. Evaluated fetal birth weight> 4000 g. In the non-cesarean section group, the extra criteria should include: nulliparous
Sampling Method: Probability Sample
Enrollment: 924 (Estimated)
Dates: Start 2022-01-30 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
vignial birth rate | up to 84 hours
  After the treatment of balloon catheter for 12 hours +oxytocin induction for up tp 72 hours, the mode of delivery will be konwn and recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Ziyan, Ph.D, Principal Investigator — Department of Obstetrics and Gynecology, First Affiliated Hospital of Nanjing Medical University
Locations (1):
- First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huisman CMA, Ten Eikelder MLG, Mast K, Oude Rengerink K, Jozwiak M, van Dunne F, Duvekot JJ, van Eyck J, Gaugler-Senden I, de Groot CJM, Franssen MTM, van Gemund N, Langenveld J, de Leeuw JW, Oude Lohuis EJ, Oudijk MA, Papatsonis D, van Pampus M, Porath M, Rombout-de Weerd S, van Roosmalen JJ, van der Salm PCM, Scheepers HCJ, Sikkema MJ, Sporken J, Stigter RH, van Wijngaarden WJ, Woiski M, Mol BWJ, Bloemenkamp KWM; PROBAAT-S project group. Balloon catheter for induction of labor in women with one previous cesarean and an unfavorable cervix. Acta Obstet Gynecol Scand. 2019 Jul;98(7):920-928. doi: 10.1111/aogs.13558. Epub 2019 Mar 7. PMID 30723900
- [Background] Battarbee AN, Palatnik A, Peress DA, Grobman WA. The Association between Cervical Exam after Ripening with Foley Balloon Catheter and Outcomes of Nulliparous Labor Induction. Am J Perinatol. 2018 Aug;35(10):1001-1005. doi: 10.1055/s-0038-1635091. Epub 2018 Feb 28. PMID 29490397